CLINICAL TRIAL: NCT00587496
Title: A 30-Day Double-Masked Study to Determine the Effect of Oral Valacyclovir or Oral Valacyclovir Plus Aspirin on the Shedding of Herpes Simplex Virus DNA in the Tears and Saliva of Volunteers Without Clinical Signs of Ocular Herpetic Disease
Brief Title: 30-Day Trial of Oral Valtrex or Valtrex Plus Aspirin on Shedding of HSV DNA in Tears and Saliva of Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Herbert E Kaufman, MD, Boyd Professor Ophthalmology, Pharmacology, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6475; EY002672
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Herpes Simplex
Keywords: HSV DNA; volunteers
MeSH Terms: conditions — Herpes Simplex | interventions — Valacyclovir; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): placebo, 6 capsules per day for 30 days
  Interventions: Drug: placebo
- 2 (Experimental): 500 mg Valtrex one capsule per day plus 5 capsules of placebo per day for 30 days
  Interventions: Drug: valacyclovir hydrochloride
- 3 (Experimental): 500 mg Valtrex capsule one per day, Acetylsalicylic acid (aspirin) 325 mg capsules three per day, plus 2 placebo capsules per day for 30 days
  Interventions: Drug: valacyclovir plus aspirin

INTERVENTIONS:
Drug: valacyclovir hydrochloride — 500 mg capsule, one per day for 30 days
  Other Names: Valtrex
  Arms: 2
Drug: placebo — lactose placebo capsule, six per day for 30 days
  Arms: 1
Drug: valacyclovir plus aspirin — 500 mg valacyclovir capsule, one per day for 30 days 325 mg acetyl salicylic acid (aspirin) capsule, three per day for 30 days placebo capsule, two per day for 30 days
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether oral Valtrex alone or in combination with aspirin will reduce the shedding of herpes simplex virus DNA in the tears and saliva from volunteers with no evidence of ocular herpes infection. The secretion of virus into the tears and saliva might make people more susceptible to virus infection in the future if their immune system becomes deficient. The study will also try to determine if there is a correlation between shedding of viral DNA and herpes virus antibodies in serum and to determine if subjects are carriers of a special form of a gene in their blood cells, the presence of which may suggest the possibility of an increased susceptability to herpes and to Alzheimer's disease and heart disease.

DETAILED DESCRIPTION:
Published studies have shown that treatment with oral acyclovir reduced clinical recurrences of ocular herpetic keratitis by about 40-50 %8, and treatment with valacyclovir, a more soluble prodrug of acyclovir, reduced the risk of transmission of genital herpes9, 10, 11. For this study, we will use the dose of valacyclovir that was shown effective in reducing the risk of transmission of HSV-2.9 The dose of 325 mg aspirin three times a day was chosen based on our experience with mice and other laboratory animals12. If it is effective and well tolerated at this dose, in future studies we will attempt to use lower doses and determine if they too may be effective.

ELIGIBILITY:
Inclusion Criteria:

* either sex
* any race
* over age of 21 years

Exclusion Criteria:

* have active ocular herpetic lesion
* had ocular herpetic lesion in past 30 days
* taking systemic or oral antiviral drugs
* have taken antiviral drugs in the past 30 days
* taking aspirin or NSAIDs
* have dry eyes
* have hypersensitivity to acyclovir or valacyclovir
* have hypersensitivity of contraindication to use of aspirin
* have bleeding disorder
* have GI ulcer
* have kidney impairment
* are pregnant or nursing
* have participated in a clinical trial in the past 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Cessation of DNA shedding above the positive detection threshold | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert E Kaufman, MD, Principal Investigator — LSU Eye Center, LSU Health Sciences Center
Locations (2):
- United States (2):
  - LSU Eye Center, New Orleans, Louisiana
  - Children's Hospital, New Orleans, Louisiana

REFERENCES:
- [Background] Kaufman HE, Azcuy AM, Varnell ED, Sloop GD, Thompson HW, Hill JM. HSV-1 DNA in tears and saliva of normal adults. Invest Ophthalmol Vis Sci. 2005 Jan;46(1):241-7. doi: 10.1167/iovs.04-0614. PMID 15623779
- [Background] Lindgren KM, Douglas RG Jr, Couch RB. Significance of Herpesvirus hominis in respiratory secretions of man. N Engl J Med. 1968 Mar 7;278(10):517-23. doi: 10.1056/NEJM196803072781001. No abstract available. PMID 4295319
- [Background] Douglas RG Jr, Couch RB. A prospective study of chronic herpes simplex virus infection and recurrent herpes labialis in humans. J Immunol. 1970 Feb;104(2):289-95. No abstract available. PMID 4312871
- [Background] Scott DA, Coulter WA, Biagioni PA, O'Neill HO, Lamey PJ. Detection of herpes simplex virus type 1 shedding in the oral cavity by polymerase chain reaction and enzyme-linked immunosorbent assay at the prodromal stage of recrudescent herpes labialis. J Oral Pathol Med. 1997 Aug;26(7):305-9. doi: 10.1111/j.1600-0714.1997.tb00220.x. PMID 9250929
- [Background] Hobson A, Wald A, Wright N, Corey L. Evaluation of a quantitative competitive PCR assay for measuring herpes simplex virus DNA content in genital tract secretions. J Clin Microbiol. 1997 Mar;35(3):548-52. doi: 10.1128/jcm.35.3.548-552.1997. PMID 9041386
- [Background] Ryncarz AJ, Goddard J, Wald A, Huang ML, Roizman B, Corey L. Development of a high-throughput quantitative assay for detecting herpes simplex virus DNA in clinical samples. J Clin Microbiol. 1999 Jun;37(6):1941-7. doi: 10.1128/JCM.37.6.1941-1947.1999. PMID 10325351
- [Background] Kessler HH, Muhlbauer G, Rinner B, Stelzl E, Berger A, Dorr HW, Santner B, Marth E, Rabenau H. Detection of Herpes simplex virus DNA by real-time PCR. J Clin Microbiol. 2000 Jul;38(7):2638-42. doi: 10.1128/JCM.38.7.2638-2642.2000. PMID 10878056
- [Background] Acyclovir for the prevention of recurrent herpes simplex virus eye disease. Herpetic Eye Disease Study Group. N Engl J Med. 1998 Jul 30;339(5):300-6. doi: 10.1056/NEJM199807303390503. PMID 9696640
- [Background] Corey L, Wald A, Patel R, Sacks SL, Tyring SK, Warren T, Douglas JM Jr, Paavonen J, Morrow RA, Beutner KR, Stratchounsky LS, Mertz G, Keene ON, Watson HA, Tait D, Vargas-Cortes M; Valacyclovir HSV Transmission Study Group. Once-daily valacyclovir to reduce the risk of transmission of genital herpes. N Engl J Med. 2004 Jan 1;350(1):11-20. doi: 10.1056/NEJMoa035144. PMID 14702423
- [Background] Crumpacker CS. Use of antiviral drugs to prevent herpesvirus transmission. N Engl J Med. 2004 Jan 1;350(1):67-8. doi: 10.1056/NEJMe038189. No abstract available. PMID 14702430
- [Background] Gebhardt BM, Varnell ED, Kaufman HE. Acetylsalicylic acid reduces viral shedding induced by thermal stress. Curr Eye Res. 2004 Aug-Sep;29(2-3):119-25. doi: 10.1080/02713680490504588. PMID 15512958
- [Background] Anon. New indications. Valtrex. FDA Drug Approvals 38:572-573, 2003.
- [Background] Sheskin DJ. Handbook of Parametric and Nonparametric tatistical Procedures. 2nd Edition. Chapman & Hall/CRC, Boca Raton, FL pp. 982,2000.